CLINICAL TRIAL: NCT06081387
Title: The Effect of Aerobic and Resistance Training in Patients With Type 2 Diabetes on Vitamin D Treatment: the DIAVITEX Project
Brief Title: The Effect of Aerobic and Resistance Training in Patients With Type 2 Diabetes on Vitamin D Treatment
Acronym: DIAVITEX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Ramon Llull (Other)
Collaborators: University of Barcelona (Other); Islamic Azad University, Sanandaj (Other); Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other); Institut Català de la Salut (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DIAVITEX-1.9
Record Dates: First submitted 2023-07-06; First posted 2023-10-13 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Vitamin D; Aerobic training; Resistance training; Insulin resistance
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Resistance Training; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Vitamin D treatment and training (Experimental): Subjects are type 2 diabetic patients on vitamin D treatment that will recieve a sarcoplasma stimulating training program. This program will run for 16 weeks and three sessions a week. This exercise plan is designed in three 5-week periods and a familiarization week session. In the first intervention week, the movements are as follows: 4 sets of eight repetitions with 20 seconds interval of rest between sets will be performed, with 60% of maximum repetitions. In the second week, with increasing intensity, the exercise will be performed with 60% 1RM. The third week, each movement will be performed in 5 sets with 6 repetitions with 20 seconds of rest between Hursts as an interval with 60% of maximum repetitions.
  Interventions: Other: Resistance training
- No vitamin D and training (Active Comparator): This will include type 2 diabetic patients not being treated with vitamin D. Sarcoplasm stimulating training system will be performed. This program will run for 16 weeks and three sessions a week. This exercise plan is designed in three 5-week periods plus a familiarization session. In the first week of intervention, the movements are as follows: 4 sets of eight repetitions with 20 seconds interval of rest between sets will be performed, with 60% of maximum repetitions. In the second week, with increasing intensity, the exercise will be performed with 60% 1RM. The third week, each movement will be performed in 5 sets with 6 repetitions with 20 seconds of rest between Hursts as an interval with 60% of maximum repetitions.
  Interventions: Other: Resistance training
- Vitamin D treatment and no traininig (No Intervention): Subjects are type 2 diabetic patients on vitamin D treatment. In this group, no exercise program will be performed.
- No Vitamin D and no training (No Intervention): Subjects are type 2 diabetic patients with no vitamin D treatment and no exericse program

INTERVENTIONS:
Other: Resistance training — Sarcoplasm stimulating training system. This program will run for a total of 16 weeks and three sessions a week. This exercise plan is designed in three 5-week periods plus a familiarization session.
  Other Names: Sarcoplasm stimulating training system, exercise.
  Arms: No vitamin D and training; Vitamin D treatment and training

SUMMARY:
The purpose of this study protocol is to assess the effect of concurrent aerobic and resistance training in patients with type 2 diabetes on vitamin D treatment

DETAILED DESCRIPTION:
Aerobic and resistance training can effectively improve clinical management in people with type 2 diabetes (T2D), leading to improvements in various health parameters, including cardiovascular health, insulin sensitivity, and muscle mass. Low vitamin D (VitD) levels are associated with T2D risk and metabolic disturbances, and some studies suggest that VitD may help reduce this risk, particularly in individuals with low VitD levels. In this line, it is widely recognized that many individuals with T2D, who may also be elderly or have osteoporosis, regularly include vitamin D treatment in their healthcare routines. Although the impact of exercise has been extensively studied, its effect on diabetic patients taking vitamin D remains inconclusive due to limited and inconsistent research findings. The aim of this study is to investigate the effect of aerobic and resistance training on clinical parameters in patients with T2D already taking VitD. The DIAVITEX study is a double-blind randomized clinical trial, including 80 individuals of both sexes (female, male) with a confirmed diagnosis of T2D and on a VitD treatment where a combination of exercises will be performed. Patients will be selected at the Primary Care Centers assigned for the study and randomly assigned to four groups: 1-Training-VitD (n=20); 2- Training (n=20), 3- VitD (n=20) and 4- No VitD (n=20). In this study, a sarcoplasm stimulating training program will be carried out online, three sessions per week for a total of 16 weeks. Before and after the physical activity subjects will perform fitness tests, as well as analysis of glycated hemoglobin, insulin resistance, lipid profile and blood inflammatory biomarkers. Nutritional education programs based on the Spanish Society of Diabetes will be provided to all participants to normalize their diets for study consistency. Expected improvements in insulin resistance, glycated hemoglobin, lipid profile, and inflammatory markers are anticipated following a 16-week regimen of exercise in patients with T2D on VitD.

ELIGIBILITY:
Inclusion Criteria:

* Adults (females or males) older than 18 years old with a diagnosis of T2D in the clinic database
* Patients who have been taking the combination therapy of metformin + sodium-glucose transport protein 2 inhibitors (iSGLT2), as recommended by the redGDPS 2023, with stable medication for the past 6 months.
* Diabetic patients taking prescribed VitD treatment for at least 6 months (intervention group) and diabetic patients not taking prescribed VitD (control group)
* Patients who signed the informed consent
* Patients capable of performing mild to moderate physical activity (to walk steadily and independently for at least 6 minutes)

Exclusion Criteria:

* Patients taking other medication different than metformin + iSGLT2 (including combinations and insulin)
* Patients taking polyvitaminic supplementation at the inclusion for at least, 1 month before the intervention
* Female subjects who are pregnant
* Patients who did not sign the informed consent

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Homeostatic Model Assessment of Insulin Resistance (HOMA IR) | Beginning of the study and after 4 months
  HOMA-IR index will be calculated by using formula (HOMA-IR=fasting glucose in mmol/l*fasting insulin in μU/ml/22.5) to determine insulin resistance
Change in Homeostasis model assessment of β-cell function (HOMA-β) | Beginning of the study and after 4 months
  The HOMA-B index will be used to quantify the pancreatic beta cells function (HOMA-B360 x fasting insulin (μU/mL) / (fasting glucose (mg/dL) - 63)).
Change in serum levels of Hemoglobin A1c. | Beginning of the study and after 4 months
  Serum levels of hemoglobin A1c will be tested in the laboratory from blood draws conducted at initial visit from a fasting blood sample.
Change in serum lipid profile | Beginning of the study and after 4 months
  Total cholesterol and High-density lipoprotein (HDL) cholesterol and triglyceride levels (mg/dL). Analysis ill be performed by the fully automatic Mindray BS380 using photometry-fixed time and point turbidimetry.
Change in weight | Beginning of the study and after 4 months
  Anthropometric measurements (weight in kilograms)
Change in waist circumference | Beginning of the study and after 4 months
  Anthropometric measurements (waist circumference in centimetre)
Change in Body Mass Index (BMI) | Beginning of the study and after 4 months
  (BMI [weight and height will be combined to report BMI] in kg/m2
Vitamin D | Beginning of the study
  Determination of Vitamin D levels in blood (ng/mL)
Vitamin D | End of the study (4 Months)
  Determination of Vitamin D levels in blood (ng/mL)

SECONDARY OUTCOMES:
Sociodemographic data | Beginning of the study
  Sociodemographic data (age, sex, ethnicity, occupation, employment status, education level, household income, alcohol intake, smoking status, current medications, family medical history, current medications taken) via questionnaire. Additionally, participants may be required to list answers to the questions e.g. list any current medications taken or age. This will all be measured in the baseline case report form.
Activity degree | Beginning of the study
  To evaluate the degree of activity, the International Physical Activity Questionnaire (IPAQ) will be administered to measure the physical activity, which through an interview assessing different items will allow to obtain the usual physical activity, being able to classify individuals in sedentary, moderate sedentary or active lifestyles.
  The IPAQ questionnaires quantifies the activity: "walk", "activities of moderate intensity" and "vigorous intensity activities" assigned to each activity about energy requirements defined in metabolic equivalent tasks (METs), being multiples of the rate of metabolic rate equivalent to kilocalories for a 60 kg.
Activity degree | End of the study (4 Months)
  To evaluate the degree of activity, the International Physical Activity Questionnaire (IPAQ) will be administered to measure the physical activity, which through an interview assessing different items will allow to obtain the usual physical activity, being able to classify individuals in sedentary, moderate sedentary or active lifestyles.
  The IPAQ questionnaires quantifies the activity: "walk", "activities of moderate intensity" and "vigorous intensity activities" assigned to each activity about energy requirements defined in metabolic equivalent tasks (METs), being multiples of the rate of metabolic rate equivalent to kilocalories for a 60 kg.
Psychological Well-being | Beginning of the study
  The psychological subjective welfare will be measured through the Psychological Well-being Index, which refers to happiness or well-being.
  A 42-item self-rating scale, which includes six dimensions: self-acceptance, positive relations with others, autonomy, environmental mastery, purpose in life and personal growth. The respondents are asked to indicate on a 6-likert scale the extent to which they agree with each statement. Each dimension may range from 7-42, with higher scores indicating greater psychological well-being.
Psychological Well-being | End of the study (4 Months)
  The psychological subjective welfare will be measured through the Psychological Well-being Index, which refers to happiness or well-being.
  A 42-item self-rating scale, which includes six dimensions: self-acceptance, positive relations with others, autonomy, environmental mastery, purpose in life and personal growth. The respondents are asked to indicate on a 6-likert scale the extent to which they agree with each statement. Each dimension may range from 7-42, with higher scores indicating greater psychological well-being.
Food consumption and adherence to the Mediterranean diet | Beginning of the study
  A 14-item questionnaire designed to assess adherence to the traditional Mediterranean Diet will be administered. Values of 0 or 1 are assigned to each item, the maximum adherence to the Mediterranean Diet is indicated by a 14-point score. A validated food frequency questionnaire with 140 items will also be administered
Food consumption and adherence to the Mediterranean diet | End of the study (4 Months)
  A 14-item questionnaire designed to assess adherence to the traditional Mediterranean Diet will be administered. Values of 0 or 1 are assigned to each item, the maximum adherence to the Mediterranean Diet is indicated by a 14-point score. A validated food frequency questionnaire with 140 items will also be administered

CONTACTS AND LOCATIONS:
Overall Officials: Joel Montane, PhD, Principal Investigator — Universitat Ramon Llull
Locations (1):
- CAP Sant Rafael, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dardashtipour E, Canivell S, Azarbayjani MA, Fuente-Vidal A, Surroca A, Gascon P, Mestres C, Anton A, Pena-Mateo MJ, Carrillo-Alvarez E, Canudas AM, Guerra-Balic M, Montane J. The effect of aerobic and resistance training in patients with type 2 diabetes on vitamin D (DIAVITEX): a study protocol. Front Public Health. 2026 Jan 5;13:1674293. doi: 10.3389/fpubh.2025.1674293. eCollection 2025. PMID 41561835